CLINICAL TRIAL: NCT02660658
Title: Optimal Single-dose Intrathecal Dexmedetomidine for Postoperative Analgesia After Lower Limb Surgery
Brief Title: Optimal Single Dose Intrathecal Dexmedetomidine for Postoperative Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R ∕ 16.01.15
Record Dates: First submitted 2016-01-16; First posted 2016-01-21 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Lower Limb Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intrathecal dexmedetomidine (Other): Up-down sequential allocation
  The dose of intrathecal DEX given to the next patient will be guided by modified Dixon's up-and-down method using 1.5 mg as a step size, which assumed to be of clinical importance
  Interventions: Drug: Intrathecal dexmedetomidine

INTERVENTIONS:
Drug: Intrathecal dexmedetomidine — The dose of intrathecal DEX given to the next patient will be guided by modified Dixon's up-and-down method using 1.5 mg as a step size, which assumed to be of clinical importance

SUMMARY:
Spinal anesthesia is a commonly used technique for lower limb surgeries offering better quality of postoperative analgesia, lower incidence of side effects, and shorter post-anesthesia care unit stay than general anesthesia. However, the relatively short duration of action of the currently available local anesthetics (LAs) make these advantages short-lived.

The risk for local anesthetic toxicity (LAST) increases with the trials to use higher concentrations or volumes of intrathecal local anesthetics to increase the duration of analgesia.

Dexmedetomidine has the potential to prolong the duration of perioperative analgesia without the need for using high doses of local anesthetics and hence with decreasing the potential risk of local anesthetic, but the increased likelihood adverse effects such as short term bradycardia and prolonged duration of motor block may offset these benefits.

DETAILED DESCRIPTION:
The aim of this study is to determine the optimal single-dose of intrathecal dexmedetomidine that prolongs the analgesic duration with the least possible side effects.

With the patients in the sitting position and the use of complete aseptic technique, 25G Whitacre spinal needles will be introduced through L2-L4 interspaces and after observing free flow of the CSF, a 3ml volume including bupivacaine 12.5mg in conjunction with dexmedetomidine (3 µg) will be injected in the first case, then the patient will be turned supine.

The dose of intrathecal DEX given to the next patient will be guided by modified Dixon's up-and-down method using 1.5 mg as a step size, which assumed to be of clinical importance.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class I to II.
* Patients scheduled for elective lower limb surgeries.

Exclusion Criteria:

* Morbid obese patients.
* Severe or uncompensated cardiovascular disease.
* Significant renal disease.
* Significant hepatic disease.
* Pregnancy.
* Lactating .
* Heart block.
* Bradyarrhythmias.
* Receiving adrenergic receptor antagonist medications.
* Receiving calcium channel blockers.
* Patients with pacemakers.
* Patients with implanted cardioverter defibrillator.
* Allergy to the study medications.
* Psychological disease.
* Neurological disorders.
* Communication barrier.
* Mental disorders.
* Epilepsy.
* Drug or alcohol abuse.
* Contraindications to spinal anaesthesia.
* Receiving opioid analgesic medications within 24 h before the operation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | For 13 hours after surgery
  The duration of analgesia, defined as the time from administering of intrathecal study solution (T0) to the time for the first rescue analgesic request

SECONDARY OUTCOMES:
Postoperative pain score | For 24 hours after surgery
  Using visual analog scale
Onset of sensory blockade | For 1 hour after initiaion of spinal anesthesia
  Onset of sensory block time defined as the time elapsed from T0 to achieve the adequate sensory level for the planned surgery.
Onset of motor blockade | For 2 hours after initiation of spinal anesthesia
  Onset of motor block time defined as the time elapsed from T0 to achieve the Bromage scale of 3
Highest dermatome level of sensory blockade | For 4 hours after initiation of spinal anesthesia
  The highest dermatome level of sensory blockade and the time needed to achieve this level from the time of injection as well as time to two segment sensory regression after T0 will be recorded
Time to motor regression | For 6 hours after initiation of spinal anesthesia
  Time to motor regression to a Bromage scale of 2
Sedation score | For 24 hours after initiation of spinal anesthesia
  Sedation scores will be assessed using a sedation scale (awake and alert= 0; quietly awake= 1; asleep but easily roused= 2; deep sleep= 3).
Postoperative nausea and vomiting | For 24 hours after initiation of spinal anesthesia
  The degree of nausea and vomiting. Nausea will be measured using a numerical rating system (none= 0; mild= 1; moderate= 2; severe= 3)
Cumulative tramadol consumption | For 24 hours after surgery
Intraoperative bradycardia | For 4 hours after initiation of spinal anesthesia
Intraoperative use of ephedrine | For 4 hours after initiation of spinal anesthesia
Intraoperative use of atropine | For 4 hours after initiation of spinal anesthesia
Intraoperative use of supplemental fentanyl | For 4 hours after initiation of spinal anesthesia
Intraoperative use of midazolam | For 4 hours after initiation of spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Samah Elkenany, MD, Principal Investigator — Lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura university, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided